CLINICAL TRIAL: NCT03227952
Title: Study of the Effectiveness of Vibrotactile Sensory Stimulation in Fibromyalgia Patients
Brief Title: Sensory Stimulation in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jesus Pujol (Other)
Responsible Party: Sponsor-Investigator, Jesus Pujol, Principal Investigator, Neurovoxel SLP
Organization: Neurovoxel SLP (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOT6932
Record Dates: First submitted 2017-07-18; First posted 2017-07-24 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a sham device identical to the active device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): Vibrotactile sensory stimulation
  Interventions: Device: Vibrotactile stimulation
- Sham (Sham Comparator): Identical device. No vibration
  Interventions: Device: Vibrotactile stimulation

INTERVENTIONS:
Device: Vibrotactile stimulation — Vibrotactile sensory stimulation will consist on whole-body stimulation with mechanical stimuli of pallesthetic type at high rate (20-90 Hz), low intensity and long daily duration (3h).

SUMMARY:
The purpose of this study is to investigate the effectiveness of low-intensity and prolonged vibrotactile sensory stimulation on symptom relieve in fibromyalgia patients.

DETAILED DESCRIPTION:
The trial will last up to 8 weeks for each subject and includes:

Three weeks treatment 1 (sham or actual) Two week washout Three weeks treatment 2 (sham or actual) Vibrotactile sensory stimulation will consist on whole-body stimulation with mechanical stimuli of pallesthetic type at high rate, low intensity and long daily duration.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of fibromyalgia according to the American College of Rheumatology (ACR) (Arthritis Rheum, 1990;33:160-172)
* Clinical symptoms are not a consequence of other medical disorder (although the presence of other disorders is not an exclusion criterion)
* Diagnoses established by an expert on fibromyalgia.
* Stable treatment of chronic use.
* Subject demonstrates an understanding of the study and a willingness to participate as evidenced by voluntary written informed consent.

Exclusion Criteria:

* Generalized inflammatory articular or rheumatic disease.
* Heavily exercise for 12 hours prior to fMRI assessment
* Severe, non-stable medical, endocrinological or neurological disorder.
* Psychotic disorder or drug abuse.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
101-point verbal rating scale (VRS) | 3 weeks
  Change on fibromyalgia key symptoms rated using 101-point verbal rating scale (combining pain, fatigue and subjective cognitive problems).

SECONDARY OUTCOMES:
Associated symptom improvement | 3 weeks
  Change on fibromyalgia secondary symptoms (including sleep disturbance, anxiety, mood, activity limitation, treatment reduction and general health rating).

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Pujol, MD, Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pujol J, Ramos-Lopez D, Blanco-Hinojo L, Pujol G, Ortiz H, Martinez-Vilavella G, Blanch J, Monfort J, Deus J. Testing the effects of gentle vibrotactile stimulation on symptom relief in fibromyalgia. Arthritis Res Ther. 2019 Jun 14;21(1):148. doi: 10.1186/s13075-019-1932-9. PMID 31200775